CLINICAL TRIAL: NCT01119690
Title: Hämeenlinna Metabolic Syndrome Research Program (HMS): Effects of Dietary Cold-pressed Turnip Rapeseed Oil and Milk Fat on Serum Lipids, Oxidized LDL, Arterial Elasticity and Platelet Function
Brief Title: Hämeenlinna Metabolic Syndrome Research Program: Effects of Rapeseed Oil on Serum Lipids and Platelet Function
Acronym: HMS-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanta-Häme Central Hospital (Other Government)
Collaborators: Linnan Klinikka Oy (Other); MTT Agrifood Research Finland (Unknown); Finnish Red Cross Blood Service (Other)
Responsible Party: Ari Palomäki, MD PhD, Head of department, Central Hospital of Kanta-Häme
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KHMetS-03-AP; HMS-03 (Other: Ethics Committee)
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Metabolic Syndrome
Keywords: Dietary; Cross-Over Study; Lipids; Rapeseed oil; Butter; Milk Fat; Unsaturated Fat; Saturated Fat; Oxidized LDL; Platelet Function; Arterial Elasticity
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapeseed oil (Active Comparator)
  Interventions: Dietary Supplement: Cold-pressed turnip rapeseed oil (CTPRO)
- Milk fat (Active Comparator)
  Interventions: Dietary Supplement: milk fat

INTERVENTIONS:
Dietary Supplement: Cold-pressed turnip rapeseed oil (CTPRO) — 1. In the dietary period of 6 to 8 weeks: CTPRO 37 ml/day.
  2. In the 5-hour oral glucose and fat tolerance test: glucose and CTPRO.
  Other Names: Virgino
  Arms: Rapeseed oil
Dietary Supplement: milk fat — 1. In dietary period of 6 to 8 weeks: 37.5 grams of butter.
  2. In the 5-hour oral glucose and fat tolerance test: glucose and cream
  Other Names: Valio butter
  Arms: Milk fat

SUMMARY:
In this study, the effects of dietary intake of cold-pressed turnip rapeseed oil (CTPRO) and milk fat are compared in men with metabolic syndrome having already participated in HMS-02 study.

DETAILED DESCRIPTION:
This open and balanced cross-over study consists of two dietary treatment phases (either Virgino (R) CTPRO or butter) for 6 to 8 weeks. They are separated from each other with an eight-week washout period. At the end of both periods and 12-hour fasting an oral glucose-fat tolerance test is carried out. Except glucose, the test consists cream (after the butter phase) and CTPRO (after the CTPRO phase).

Otherwise, the subjects (n=43) are asked to maintain their normal dietary habits.

ELIGIBILITY:
Inclusion Criteria:

* 43 men with metabolic syndrome having already participated in the HMS-02 Study
* Willing to participate in a demanding dietary study

Exclusion Criteria:

Ages: 31 Years to 66 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-09; Primary Completion 2005-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Circulating lipids | 6 to 8 weeks
  At the end of both 6- to 8-week dietary periods, fasting values of circulating lipids including oxidized LDL are determined
Platelet function | 6 to 8 weeks
  At the end of both 6- to 8-week dietary periods, platelet function is determined
Glucose tolerance | 5 hours
  During a 5-hour oral glucose-fat tolerance test the area under curve of plasma glucose and insulin concentration is determined

SECONDARY OUTCOMES:
Arterial elasticity | 6 to 8 weeks
  At the end of both 6- to 8-week dietary periods, arterial elasticity is determined
Serum triglyceride AUC | 5 hours
  During a 5-hour oral glucose-fat tolerance test the area under curve of serum triglyceride concentration is determined
Platelet function | 5 hours
  During a 5-hour oral glucose-fat tolerance test the platelet function is determined

CONTACTS AND LOCATIONS:
Overall Officials: Ari K Palomäki, MD PhD, Study Director — Central Hospital of Kanta-Häme; Kalevi Oksanen, MD PhD, Study Director — Central Hospital of Kanta-Häme
Locations (4):
- Finland (4):
  - Linnan Klinikka, Hämeenlinna
  - Central Hospital of Kanta-Häme, Hämeenlinna
  - Finnish Red Cross Blood Transfusion Service, Helsinki
  - MTT Agrifood Research Finland, Jokioinen

REFERENCES:
- [Derived] Saarinen HJ, Husgafvel S, Pohjantahti-Maaroos H, Wallenius M, Palomaki A. Improved insulin sensitivity and lower postprandial triglyceride concentrations after cold-pressed turnip rapeseed oil compared to cream in patients with metabolic syndrome. Diabetol Metab Syndr. 2018 May 4;10:38. doi: 10.1186/s13098-018-0340-7. eCollection 2018. PMID 29755591
- [Derived] Saarinen HJ, Sittiwet C, Simonen P, Nissinen MJ, Stenman UH, Gylling H, Palomaki A. Determining the mechanisms of dietary turnip rapeseed oil on cholesterol metabolism in men with metabolic syndrome. J Investig Med. 2018 Jan;66(1):11-16. doi: 10.1136/jim-2017-000495. Epub 2017 Aug 11. PMID 28801309
- [Derived] Palomaki A, Pohjantahti-Maaroos H, Wallenius M, Kankkunen P, Aro H, Husgafvel S, Pihlava JM, Oksanen K. Effects of dietary cold-pressed turnip rapeseed oil and butter on serum lipids, oxidized LDL and arterial elasticity in men with metabolic syndrome. Lipids Health Dis. 2010 Dec 1;9:137. doi: 10.1186/1476-511X-9-137. PMID 21122147